CLINICAL TRIAL: NCT05011825
Title: A Pilot Evaluation of the Pregnant Moms' Empowerment Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Notre Dame (Other)
Collaborators: University of Memphis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 17-08-4035
Record Dates: First submitted 2021-08-02; First posted 2021-08-18 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-11

CONDITIONS: Violence; Depression; Posttraumatic Stress Disorder; Parenting; Infant Development; Child Behavior
MeSH Terms: conditions — Depression; Stress Disorders, Post-Traumatic; Child Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pregnant Moms' Empowerment Program (Experimental): The PMEP is a 5-session program, delivered prenatally. The first three sessions address violence and mental health and the final two sessions address labor/delivery, infant health and early parenting.
  Interventions: Behavioral: Pregnant Moms' Empowerment Program
- Control (No Intervention): Control group participants received information about community resources, but did not receive any study-related intervention.

INTERVENTIONS:
Behavioral: Pregnant Moms' Empowerment Program — The first session introduces women to the group, seeks to build an alliance and sense of group cohesion, and provides safety planning. The second session addresses intergenerational patterns of violence and how such violence contributes to psychopathology in both the prenatal and postnatal period, focusing on violence prevention. Information regarding cognitive restructuring, behavioral activation, and coping styles is provided in session three, as well as the role of healthy relationships and social supports in promoting resilience. This session begins with discussion on health in pregnancy, labor/delivery, and coordinating care across providers. This session also provides psychoeducation related to post-delivery parenting, including infant safety, care and breastfeeding. In the final session, group leaders assist mothers with identification, sensitivity, and responsiveness to infant cues.
  Arms: Pregnant Moms' Empowerment Program

SUMMARY:
This project will use a longitudinal design with assessments at baseline (T1), post-treatment (T2), 3 month post-partum (T3), 1 year postpartum (T4) and 3.5-5 years postpartum to examine whether the PMEP improves participants': a) mental health (depression, PTSD) and resilience, b) parenting skills, c) birth, infant, and toddler developmental outcomes, and d) lowers re-victimization rates. We hypothesize significantly improved outcomes in the intervention group compared to the control group at post-treatment and at all follow-ups. The pilot will use a quasi-randomized design, with participants assigned to alternating treatment and control blocks. Analyses will be conducted using intent to treat and per protocol methods. Following group assignment, all women will be scheduled for a baseline interview at a time convenient for the participant. Participant interviews will take approximately 1.5 hours. Mothers will be compensated with a gift card in the amount of 40 USD for each interview. In addition to the core evaluation metrics, mothers' demographic information will be obtained (age, relationship status, employment, education, number of children, income). Following the baseline interview, the PMEP will be provided to the treatment group; participants will receive 2-hours of contact time per week for 5 weeks (2-hour sessions, held once weekly). Women will receive reminder calls the day of each session to identify and resolve any barriers to attendance (e.g., transportation). Taxi fare will be supported for women who are unable to obtain transportation if the bus is not feasible. Following the completion of the PMEP groups or - for the control group - after 5-6 weeks has passed, all participants will complete a second interview. This interview will include all of the core measures of hypothesized treatment change, thereby permitting a comparison between women in the treatment and control groups over time. All women will be invited in a third time when their infant is 3 months old and again when their infant is 1 year of age to evaluate parenting and infant outcomes. Women will participate in a brief phone assessment when their children are between 3.5 and 5 years of age that includes all primary study outcomes.

ELIGIBILITY:
Inclusion Criteria:

* at least 16 years of age
* experienced IPV in the past year
* currently pregnant (<33 weeks)
* English speaking

Exclusion Criteria:

* insufficient fluency in English to participate in interviews/groups

Ages: 16 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 137 (Actual)
Dates: Start 2017-03-15 (Actual); Primary Completion 2021-02-15 (Actual); Study Completion 2021-02-15 (Actual)

PRIMARY OUTCOMES:
Center for Epidemiological Studies Depression Scale | Change from baseline assessment to post-test (5-6 weeks later)
  Depression
Center for Epidemiological Studies Depression Scale | Change from baseline assessment to 3 months postpartum
  Depression
Center for Epidemiological Studies Depression Scale | Change from baseline assessment to 12 months postpartum
  Depression
Center for Epidemiological Studies Depression Scale | Change from baseline assessment to 3.5-5 years postpartum
  Depression
PTSD Checklist - 5 | Change from baseline assessment to post-test (5-6 weeks later)
  Posttraumatic Stress
PTSD Checklist - 5 | Change from baseline assessment to 3 months postpartum
  Posttraumatic Stress
PTSD Checklist - 5 | Change from baseline assessment to 12 months postpartum
  Posttraumatic Stress
PTSD Checklist - 5 | Change from baseline assessment to 3.5-5 years postpartum
  Posttraumatic Stress
Connors Davidson Resilience Scale | Change from baseline assessment to post-test (5-6 weeks later)
  Resilience
Connors Davidson Resilience Scale | Change from baseline assessment to 3 months postpartum
  Resilience
Connors Davidson Resilience Scale | Change from baseline assessment to 12 months postpartum
  Resilience
Connors Davidson Resilience Scale | Change from baseline assessment to 3.5-5 years postpartum
  Resilience
Conflict Tactics Scales - Revised | Change from baseline assessment to post-test (5-6 weeks later)
  Intimate Partner Violence
Conflict Tactics Scales - Revised | Change from baseline assessment to 3 months postpartum
  Intimate Partner Violence
Conflict Tactics Scales - Revised | Change from baseline assessment to 12 months postpartum
  Intimate Partner Violence
Conflict Tactics Scales - Revised | Change from baseline assessment to 3.5-5 years postpartum
  Intimate Partner Violence
Adult Adolescent Parenting Inventory | Change from baseline assessment to post-test (5-6 weeks later)
  Parenting Attitudes
Adult Adolescent Parenting Inventory | Change from baseline assessment to 3 months postpartum
  Parenting Attitudes
Adult Adolescent Parenting Inventory | Change from baseline assessment to 12 months postpartum
  Parenting Attitudes
Adult Adolescent Parenting Inventory | Change from baseline assessment to 3.5-5 years postpartum
  Parenting Attitudes
Karitane Parenting Inventory | Change from baseline assessment to post-test (5-6 weeks later)
  Parenting Confidence
Karitane Parenting Inventory | Change from baseline assessment to 3 months postpartum
  Parenting Confidence
Karitane Parenting Inventory | Change from baseline assessment to 12 months postpartum
  Parenting Confidence
Pregnancy Risk and Monitoring System (PRAMS) | Differences between groups at 3 months postpartum
  Labor, Delivery and Breastfeeding
Pregnancy Risk and Monitoring System (PRAMS) | Differences between groups at 12 months postpartum
  Labor, Delivery and Breastfeeding
Infant Development | Difference between groups at 12 months post partum
  Bayley Scales of Infant Development
Infant Development | Differences between groups at 3 months postpartum
  Bayley Scales of Infant Development
Infant Behavior Questionnaire | Differences between groups at 12 months post partum
  Infant Temperament
Maternal Sensitivity and Infant Affect Regulation | Differences between groups at 3 months postpartum
  Coded free play data
Maternal Sensitivity and Infant Affect Regulation | Differences between groups at 12 months postpartum
  Coded free play data

SECONDARY OUTCOMES:
Lubben Social Network Scale | Change from baseline to posttest (5-6 weeks later)
  Social Support
Lubben Social Network Scale | Change from baseline to 3 months postpartum
  Social Support
Lubben Social Network Scale | Change from baseline to posttest 12 months postpartum
  Social Support
Lubben Social Network Scale | Change from baseline to posttest 3.5-5 years postpartum
  Social Support
Rotter Locus of Control Scale | Change from baseline to post-test (5-6 weeks later)
  Locus of Control
Rotter Locus of Control Scale | Change from baseline to 3 months postpartum
  Locus of Control
Rotter Locus of Control Scale | Change from baseline to 12 months postpartum
  Locus of Control
Child behavior checklist | 3.5-5 years postpartum
  Child adjustment

OTHER OUTCOMES:
Breastfeeding Behavior Scale | Differences between groups at 12 months post partum
  Breastfeeding attitudes
Postpartum Depression Scale | 3 months postpartum
  Postpartum depression

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of NotreDame, Notre Dame, Indiana
  - University of Memphis, Memphis, Tennessee

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Howell KH, Gilliam HC, Carney JR, Maloney CA, Miller-Graff LE. Long-term effects of the Pregnant Moms' Empowerment Program (PMEP) on intimate partner violence revictimization, maternal mental health, and child internalizing and externalizing problems. J Consult Clin Psychol. 2025 Sep;93(9):642-651. doi: 10.1037/ccp0000976. PMID 40875361